CLINICAL TRIAL: NCT01925261
Title: A Randomized, Double-blind, Placebo-controlled, Multi-dose Phase 2 Study Evaluating the Safety and Efficacy of Intra-articular Injections of TPX-100 in Subjects With Mild to Moderate Patello-Femoral Osteoarthritis Involving Both Knees
Brief Title: A Study Evaluating the Safety and Efficacy of Intra-articular Injections of TPX-100 in Subjects With Mild to Moderate Patello-Femoral Osteoarthritis Involving Both Knees
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OrthoTrophix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPX-100
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2015-05

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; bilateral; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TPX-100 Cohort 1 (Placebo Comparator): Cohort 1 will be 20mg dose of TPX-100 in one randomized knee, compared to placebo treated knee
  Interventions: Drug: TPX-100 20mg; Drug: Placebo
- TPX-100 Cohort 2 (Placebo Comparator): Cohort 2 will be 50mg dose of TPX-100 in one randomized knee compared to placebo treated knee
  Interventions: Drug: TPX-100 50mg; Drug: Placebo
- TPX-100 Cohort 3 (Placebo Comparator): Cohort 3 will be 100mg dose of TPX-100 in one randomized knee compared to placebo treated knee
  Interventions: Drug: TPX-100 100mg; Drug: Placebo
- TPX-100 Cohort 4 (Placebo Comparator): Cohort 4 will be 200mg dose of TPX-100 in one randomized knee, compared to placebo treated knee
  Interventions: Drug: TPX-100 200mg; Drug: Placebo
- Part B (Placebo Comparator): Part B will be 200mg dose of TPX-100 in one randomized knee, compared to placebo treated knee
  Interventions: Drug: TPX-100 200mg; Drug: Placebo

INTERVENTIONS:
Drug: TPX-100 50mg
  Other Names: 50mg of TPX-100
  Arms: TPX-100 Cohort 2
Drug: TPX-100 100mg
  Other Names: 100mg of TPX-100
  Arms: TPX-100 Cohort 3
Drug: TPX-100 200mg
  Other Names: 200mg of TPX-100
  Arms: Part B; TPX-100 Cohort 4
Drug: TPX-100 20mg
  Other Names: 20mg of TPX-100
  Arms: TPX-100 Cohort 1
Drug: Placebo

SUMMARY:
This one-year study is designed to investigate the safety and efficacy of TPX-100, a 23-amino acid chondrogenic peptide, delivered by intra-articular injection, in regeneration of knee cartilage in subjects with bilateral osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 25 and ≤ 75
2. Patello-femoral osteoarthritis of both knees of mild to moderate severity with intact meniscus and ligamentous stability (cruciate and collateral ligaments)

   * Clinically, as determined by screening questionnaire and judgment of the Principal Investigator (may be supported by imaging studies of knees); confirmed by centrally read screening MRI of both knees indicating ICRS Grade 1-3, or ICRS Grade 4 with only focal defects, no greater than 1 cm.
   * Meniscus intact (MRI degenerative signal up to and including grade II acceptable)
   * Cruciate and collateral ligament stability as defined by clinical examination
3. Able to read, understand, sign and date the subject informed consent
4. Willingness to use only acetaminophen as the primary analgesic (pain-relieving) study medication. The maximum dose of acetaminophen must not exceed 4 grams/day (4000 mg per day).
5. Willingness to use only hydrocodone/acetaminophen for breakthrough pain during the injection period (through study day 30).
6. Willingness not to use non-steroidal anti-inflammatory drugs (NSAIDS) such as aspirin, ibuprofen, naproxen for the first 30 days of the study.
7. Female subjects of child bearing potential who are sexually active (non-abstinent) must agree to and comply with using 2 highly effective methods of birth control (oral contraceptive, implant, injectable or indwelling intrauterine device, condom with spermicide, or sexual abstinence) while participating in the study.

Exclusion Criteria:

1. Contraindication to MRI, including: metallic fragments, clips or devices in the brain, eye, or spinal canal; implanted devices that are magnetically programmed; weight > 300 lbs.; moderate or severe claustrophobia; previous intolerance of MRI procedure
2. ICRS grade greater than Grade 3, or Grade 4 focal defects greater than 1 cm, as confirmed by centrally-read screening MRI
3. MRI evidence of inflammatory or hypertrophic synovitis
4. Prior surgery in the knees, excluding procedures for debridement only (no microfracture)
5. Joint replacement or any other knee surgery planned in the next 12 months
6. History of rheumatoid arthritis, psoriatic arthritis, or any other autoimmune or infectious cause for arthritis
7. Knee effusion >2+ on the following clinical scale:

   * Zero = No wave produced on downstroke
   * Trace = Small wave on medial side with downstroke
   * 1+ = Larger bulge on medial side with downstroke
   * 2+ = Effusion spontaneously returns to medial side after upstroke (no downstroke necessary)
   * 3+ = So much fluid that it is not possible to move the effusion out of the medial aspect of the knee
8. Last viscosupplementation (e.g. Synvisc® or similar hyaluronic acid product) injected into either knee < 3 months before screening
9. Last intra-articular knee injection of corticosteroids < 2 months before screening
10. Use of any steroids (except inhaled corticosteroids for respiratory problems) during the previous month before screening
11. Known hypersensitivity to TPX-100
12. Known hypersensitivity to acetaminophen or hydrocodone
13. History of arthroscopy in either knee in the last 3 months before screening
14. History of septic arthritis, gout or pseudo-gout, of either knee in previous year before screening
15. Clinical signs of acute meniscal tear (locking, new acute mechanical symptoms consistent with meniscal tear)
16. Patellar chondrocalcinosis on X-Ray
17. Skin problem, rash or hypersensitivity, affecting either knee at the injection site
18. Bleeding problem, platelet or coagulation deficiency contraindicating, in the doctor's opinion, any intra-articular injection
19. Active systemic infection
20. Current treatment or treatment within the previous 2 years prior to the Screening Visit for any malignancy except basal cell or squamous cell carcinoma of the skin, unless with specific written permission is provided by the Sponsor's medical monitor
21. Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period
22. Participation in other clinical osteoarthritis drug studies within one year prior to screening
23. Currently taking Paclitaxel (mitotic inhibitor), and or Natalizumab (anti-integrin monoclonal antibody).
24. History of significant liver disease or consumption of more than 3 alcoholic drinks a day. (Definition of one alcoholic drink: 12-ounces of beer, 8-ounces of malt liquor, 5-ounces of wine, 1.5-ounces or a "shot" of 80-proof distilled spirits or liquor such as gin, rum, vodka, or whiskey).

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in cartilage thickness in the patello-femoral compartment as measured on standardized MRI from baseline to 12 months | 12 months
  Change in cartilage thickness in the patello-femoral compartment from baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- C3 Clinical Research Associates, Seattle, Washington, United States

REFERENCES:
- [Derived] McGuire D, Bowes M, Brett A, Segal NA, Miller M, Rosen D, Kumagai Y. Study TPX-100-5: intra-articular TPX-100 significantly delays pathological bone shape change and stabilizes cartilage in moderate to severe bilateral knee OA. Arthritis Res Ther. 2021 Sep 17;23(1):242. doi: 10.1186/s13075-021-02622-8. PMID 34535197